CLINICAL TRIAL: NCT02926079
Title: Investigation of Mechanisms for Transmission of Impaired Glucose Metabolism in Infants Exposed to Diabetes in Utero
Acronym: IMAGINE
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Leanne Redman, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2016-071
Record Dates: First submitted 2016-09-19; First posted 2016-10-06 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy; Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Maternal Blood Collection: Approximately 33mL of blood will be collected during the visit.
  Infant Blood Collection: Approximately 2mL of blood will be collected during the visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant women diagnosed with gestational diabetes
- Pregnant women with normal pregnancy

SUMMARY:
This proposed study; Investigation of mechanisms for transmission of impaired glucose metabolism in infants exposed to diabetes in utero, will test the overarching hypothesis that impaired maternal substrate oxidation (metabolic inflexibility) and placental lipotoxicity are characteristics of diabetic pregnancies and in utero development within these conditions programs a metabolically inflexible phenotype in the offspring.

DETAILED DESCRIPTION:
This translational research study will obtain paired measures of metabolic flexibility (postprandial RQ minus basal RQ) in response to a standardized meal by indirect calorimetry in mother:infant dyads of diabetic and non-diabetic pregnancies. The downstream effects of the intrauterine exposure to diabetes and gestational lipotoxicity will be tested in the infant: 1) at birth by studying adipogenic pathways and mitochondrial function in umbilical cord mesenchymal stem cells cultured in myogenic conditions[13], and 2) by studying metabolic flexibility in the infant in a whole body infant calorimeter in response to a standardized meal.

Mothers will be enrolled between (33-35 weeks of gestation) and their infants will be enrolled between 10-30 days of life with the following aims.

Aim 1. Characterize metabolic flexibility and lipotoxicity in diabetic and non-diabetic pregnancies.

Hypothesis 1A: In response to a standardized meal in late pregnancy, diabetic pregnancies will be metabolically inflexible (blunted switch in RQ from the fasted state to the postprandial state) compared to non-diabetic pregnancies matched for maternal age and pregravid BMI.

Hypothesis 1B: Placenta from diabetic pregnancies will have higher lipid content, reduced mitochondrial content and lower rates of mitochondrial oxygen consumption compared to placenta from non-diabetic pregnancies.

Aim 2. Test whether intrauterine exposure to maternal diabetes infers disordered substrate oxidation in offspring at birth (in myocytes cultured from umbilical cord mesenchymal stem cells) and early in postnatal life (metabolic flexibility in response to a standardized meal).

Hypothesis 2A: Umbilical cord mesenchymal stem cells cultured in myogenic conditions from diabetic pregnancies will have greater lipid content, reduced mitochondrial content, and lower rates of mitochondrial electron transport oxygen consumption and fatty acid oxidation.

Hypothesis 2B: In response to a standardized meal, offspring of diabetic pregnancies will be metabolically inflexible (blunted switch in RQ from the pre- to postprandial state) compared to offspring of non-diabetic pregnancies.

ELIGIBILITY:
Inclusion Criteria (Mother):

* BMI between 20 kg/m2 and 40 kg/m2 prior to the current pregnancy (determined by self-report and confirmation of pregravid BMI of the index pregnancy from the prenatal record)
* Completion of standardized glucose tolerance testing (between 24-28 weeks gestation) in the index pregnancy; either a single 2 hour, 75g glucose tolerance test or the two-step: 1 hour 50g and 3 hour 100g glucose tolerance test to confirm diagnosis of gestational diabetes mellitus or normal glucose tolerance
* Medically cleared for participation in the study by primary care obstetrician or midwife
* Medically cleared for participation by the Medical Investigator
* Medical record release (prenatal record, hospital delivery record) for study staff to access information in the medical record related to the current and if applicable, the prior pregnancy.
* Willingness to enroll the infant in the study provided inclusion/exclusion criteria pertaining to the infant are met

Inclusion criteria (Infant):

* Born full-term (>37,0 weeks gestation)
* Available for clinical assessments between 10-30 days old
* Healthy

Exclusion Criteria (Mother):

* Use of insulin therapy in the index pregnancy
* History of preterm birth
* History of intrauterine growth-restriction
* Evidence of gestational hypertension (SBP >160 mmHg & DBP >110 mmHg)
* HIV or AIDS (self-reported)
* Planned termination of pregnancy or adoption or unwillingness to enroll the infant in the study

Exclusion Criteria (Infant):

* Using medications to treat a chronic condition (does not include use of vitamin supplements or PRN medication for flatulence)
* Unwilling or unable to be fed 2 fl oz of infant formula
* Diagnosed with a congenital abnormality or disability that would render testing unsafe or would interfere with data collection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Up to 20 pregnant women with and without gestational diabetes mellitus with a BMI between 20 kg/m2 and 40 kg/m2 prior to the current pregnancy.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Metabolic flexibility - Mother | One day
  Assessed during a mixed-meal test as the difference in RQ between the postprandial period and the fasting period via indirect calorimetry.

SECONDARY OUTCOMES:
Metabolic Flexibility - Infant | One day
  Assessed during a standard infant formula test as the difference in RQ between the postprandial and the fasting period via indirect calorimetry.
Lipid content in placenta samples | One day (delivery)
  Lipid content will be measured in placenta samples via immunohistochemistry antibody staining for lipid droplet proteins and by Oil Red O staining.
Mitochondrial oxygen consumption rates in placenta samples | One day (delivery)
  Oxygen consumption rates of isolated mitochondria from placenta will be measured by the SeaHorse device.
Fat content in umbilical cord mesenchymal stem cells | One day (delivery)
  Mesenchymal stem cells will be differentiated to a myogenic state and assessed for lipid content via Oil Red O staining
Oxygen consumption rates in umbilical cord mesenchymal stem cells | One day (delivery)
  Mesenchymal stem cells will be differentiated to a myogenic state and assessed for oxygen consumption rates using the Oroboros device.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided